CLINICAL TRIAL: NCT06667882
Title: Safe Delivery of Thrombolytic Treatment for Pulmonary Embolism Using ClotPro® Viscoelastic Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Janos Fazakas MD, PhD, Associate Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65187-5/2021/EÜIG
Record Dates: First submitted 2024-10-24; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Embolism Subacute Massive; Complication of Treatment; Fibrinolysis; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional thrombolysis group (Active Comparator): A fixed dose of rtPA will be delivered, preferably with coagulation monitoring. The rtPA dose is 0.6 mg/kg over 15 minutes (with a maximum dose of 50 mg) for circulatory collapse, and 100 mg over 2 hours for circulatory instability that persists despite circulatory support
  Interventions: Drug: Alteplase Injectable Product
- ClotPro-controlled variable dose of thrombolytic treatment. (Experimental): A variable dose will be delivered, according to ClotPro EX, IN, AP, FIB, ECA, RVV, TPA results. The starting rtPA dose is 0.15-0.04 mg/kg in bolus, the starting maintaining dose for the first lysis hour the same. ClotPro tests is made in every 1 h treatment. The maintaining rtPA dose if it is needed, will be increased, till EX, IN, ECA efficient lysis could be detected. On the other hand the reduction of the maintaining dose was permitted based on FIB MCF alarming decline. The thrombolysis treatment is stopped if the circulatory instability and/or circulatory support ceased. Based on FIB MCF results fibrinogen concentrate coadministration on safety reason is permitted.
  Interventions: Drug: Alteplase Injectable Product

INTERVENTIONS:
Drug: Alteplase Injectable Product — The 2019 ESC guideline for the diagnosis and management of acute pulmonary embolism (PE) recommended thrombolytic therapy only in high-risk PE cases because of the bleeding risk. The most often used drug for thrombolysis is the rtPA and the recommended dose is 100 mg over two hours. According to the literature, the risk of major haemorrhage is 10-13% and fatal or intracranial bleeding is 1.7-3.6% among patients receiving thrombolysis.

SUMMARY:
The aim of this work was to reduce the bleeding risk during thrombolysis using the viscoelastic blood coagulation tests.

DETAILED DESCRIPTION:
Patient data The patients' age, body measurements, general and coagulation-related medical history, SARS-COV2 status, APACHE-II, frailty score will be recorded.

Sampling times and examinations

The following considerations will be taken into account in the course of examining and providing care to the patients:

Imaging procedures:

CT angiography of the chest To confirm embolism and the results of lysis 12 to 24 hours after it is completed mandatory Echocardiography Right ventricle diameter mandatory views to be recorded: TAPSE mandatory parasternal longitudinal section IVC minimum and maximum diameter mandatory parasternal basal cross-section extent of tricuspid regurgitation mandatory apical 4 chamber estimated APsys mandatory subcostal 4 chamber D sign? mandatory IVC McConnel sign? optional 60/60 sign optional right heart thrombus optional Tricuspid annulus with reduced S' (<9.5 cm/s) tissue doppler optional Lower limb Doppler ultrasound Search for the origin of thromboembolism, preferably prior to lysis optional Table 2: Summary of the imaging procedures required for the study The condition for enrolment into the study is PE confirmed by CT angiography of the chest, with haemodynamic impact confirmed by echocardiography; the recording of the test in the IMPAX system is also a requirement. To assess the effectiveness of thrombolysis, echocardiography must be repeated after the lysis is completed, and then 12 to 24 hours later; the same is true for long-term follow-up.

Blood analyses:

Laboratory tests blood type + antibody screening mandatory blood count mandatory INR mandatory aPTI mandatory D-dimer mandatory fibrinogen mandatory Troponin T mandatory NT-proBNP mandatory creatinine mandatory urea mandatory electrolytes (Na+; K+; Ca2+ (t/ion); Mg2+; Cl-, phosphate) mandatory liver function (AST, ALT, LDH) mandatory Blood gases pH; pO2; pCO2 mandatory HCO3-; BE mandatory hgb mandatory Na+; K+; Ca2+; Cl- mandatory blood glucose mandatory lactate mandatory

Table 3: Summary of the laboratory and point-of-care blood tests required for the study The above lab parameters are planned to be obtained upon enrolment of a patient. Also, in addition to regular blood gas testing during the treatment, targeted testing for coagulation parameters and factors might be necessary.

Invasive interventions:

Arterial cannulation invasive pressure monitoring; pressurised infusion without heparin! mandatory PVC at least one, but preferably two, minimum G18 mandatory CVC only if vasopressor must be delivered; giving dobutamine to increase inotropy is not in itself an indication for a CVC! optional bladder catheter indication should be considered; if in doubt, should be inserted before the start of lysis optional endotracheal tube only for an indication not associated with pulmonary embolism optional Table 4: Considerations for the invasive interventions required for the study

Study phase and follow-up The study period is expected to last from 1 October 2021 to 31 December 2024. Follow-up (subject to a separate consent from the patients) will take place 1, 3 and 12 months after the thrombolysis and is planned to include quality of life questionnaires (EuroQOL -5D-5L), assessment of physical capacity (6MW, or, if unfeasible, Timed Up&Go test), echocardiography, ClotPro and blood gas testing.

Methodology and organisation of the study Potential recruits are the patients of Semmelweis University with relevant impact on circulation (high-risk or intermediate to high-risk categories), whose PE is confirmed by CT angiography of the chest. Patients may come from the Emergency Care Unit or may be hospitalised patients from another department. The patient will then be admitted to the Anaesthesiology and Intensive Therapy Clinic and receive care there until stabilised.

Instable patients who are enrolled will all be administered a fixed dose (100 mg/h) (see the section 'Inclusion criteria'). High risk or intermediate-high risk patients who can be stabilised will be randomised and then receive either a fixed dose (100 mg/2h) or a ClotPro-controlled variable dose of thrombolytic treatment.

Coagulation tests

ClotPro tests are planned before and regularly after the start of treatment: EX, IN, FIB, TPA, AP, RVV and ECA tests will be required.

Statistical methods Statistical analyses will be performed by Social Sciences software (SPSS; SPSS Inc, Chicago, Illinois, USA).

Continuous and discrete variables will be analysed by independent samples t tests (two categories) and one-way analyses of variance (one-way ANOVA; more categories), respectively. Two continuous variables will be compared by Spearman's rank correlation test. Discrete variables will be tested by Pearson's Chi squared test. Ordinary variables will be compared by Mann-Whitney U test or Kruskal-Wallis test. For multivariate analyses, logistic regression models will be generated.

Significance level will be set to 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary embolism confirmed by CT angiography of the chest, and planned systemic thrombolysis, taking into account the following:
* For indications based on circulatory collapse or circulatory instability that persists despite circulatory support, a fixed dose will be delivered, preferably with coagulation monitoring. The rtPA dose is 0.6 mg/kg over 15 minutes (with a maximum dose of 50 mg) for circulatory collapse, and 100 mg over 2 hours for circulatory instability that persists despite circulatory support.
* Otherwise, a regime relevant to our study is followed in the following cases in the individuals randomised to the study treatment group:
* Haemodynamic instability resolved through inotropic and/or vasopressor therapy, or
* In the event of right heart strain confirmed by echocardiography, and elevated cardiac biomarker (hs Troponin-T/NT-proBNP) in a haemodynamically stable patient, the regime to be followed will be determined by the monitoring results.

Exclusion criteria:

* Failure to obtain informed consent from the patient (or from the closest relative of an incapacitated patient).
* Coagulation tests included in the study protocol cannot be performed for any technical reason or samples cannot be collected.
* Patients <18 years of age at the onset of pulmonary embolism.
* Pregnancy.
* The following risk factors are known or currently present in the patient:

  * Haemorrhagic stroke at any time in the medical history
  * Major trauma or head injury within the last three weeks
  * Incorrigible bleeding abnormality
  * Active bleeding that cannot be attenuated
  * Therapy refractory hypertension
  * Infective endocarditis
* Patients lacking legal competence and the guardian or closest relative cannot be contacted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Major, life threatening bleeding due to profuse bleeding | during the treatment with tPA (on the control arm 2 hours, on the intervention arm variable > 2 hours)
  Hemorrhagic shock due to profuse bleeding:
  * hemoglobin reduction > 30 g/l AND
  * Systolic blood pressure < 90 mmHg OR
  * Reduction in systolic blood pressure > 40 mmHg OR
  * Preserved systolic blood pressure achieved through increased dose of inotropic/vasopressor therapy
Major, life threatening bleeding due to intracranial haemorrhage | during the treatment with tPA (on the control arm 2 hours, on the intervention arm variable > 2 hours)
  Intracranial hemorrhage - new onset of neurological symptoms
Minor bleeding: Haemoglobin reduction > 10g/l during the treatment | during the treatment with tPA (on the control arm 2 hours, on the intervention arm variable > 2 hours)
  Haemoglobin reduction > 10g/l, but less, than 30 g/l

SECONDARY OUTCOMES:
Efficiency - Short therm: hemodynamic stabilization | 36 hours after treatment
  absence of circulatory shock/circulatory support ceased
Efficiency - Short therm: significant regression or absence of embolus mass on post treatment pulmonary angio CT scan | 24 hours after treatment
Efficiency - Long therm: further improvement on pulmonary CT scan | One month after the treatment
  Long term: further improvement on pulmonary CT scan
Efficiency - Long therm: absence of right hearth failure on echocardiography | One year after the treatment
  Absence of right heart failure on echocardiography:
  * no D-sign AND
  * basal right ventricle/left ventricle ratio < 1 AND
  * tricuspidal annular plain systolic excursion > 16 mm AND
  * Tissue Doppler Imaging: peak systolic velocity of tricuspid annulus > 9.5 cm/s
Efficiency - Long therm: improvement on 6 minutes walking test | One year after the treatment
  Long term: improvement on 6 minutes walking test. The measured parameters:
  * 6 minutes walking test distance ( 6MWD - in meter)
  * 6MWD/predicted 6MWD (%)
  * distance desaturation product (DSP - m%)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Anesthesiology and Intensive Therapy, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zatroch I, Dinya E, Fazakas J. New under the sun: ClotPro's ECA-test detects hyperfibrinolysis in a higher number of patients, more frequently and 9 min earlier. Blood Coagul Fibrinolysis. 2023 Mar 1;34(2):99-104. doi: 10.1097/MBC.0000000000001185. Epub 2022 Dec 15. PMID 36519572
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Background] Weinstein T, Deshwal H, Brosnahan SB. Advanced management of intermediate-high risk pulmonary embolism. Crit Care. 2021 Aug 31;25(1):311. doi: 10.1186/s13054-021-03679-2. PMID 34461959
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Meneveau N, Seronde MF, Blonde MC, Legalery P, Didier-Petit K, Briand F, Caulfield F, Schiele F, Bernard Y, Bassand JP. Management of unsuccessful thrombolysis in acute massive pulmonary embolism. Chest. 2006 Apr;129(4):1043-50. doi: 10.1378/chest.129.4.1043. PMID 16608956
- [Background] Hoffman M. A cell-based model of coagulation and the role of factor VIIa. Blood Rev. 2003 Sep;17 Suppl 1:S1-5. doi: 10.1016/s0268-960x(03)90000-2. PMID 14697207
- [Background] Zatroch I, Smudla A, Babik B, Tanczos K, Kobori L, Szabo Z, Fazakas J. [Procoagulation, hypercoagulation and fibrinolytic "shut down" detected with ClotPro(R) viscoelastic tests in COVID-19 patients]. Orv Hetil. 2020 May;161(22):899-907. doi: 10.1556/650.2020.31870. Hungarian. PMID 32453702
- [Background] Bachler M, Bosch J, Sturzel DP, Hell T, Giebl A, Strohle M, Klein SJ, Schafer V, Lehner GF, Joannidis M, Thome C, Fries D. Impaired fibrinolysis in critically ill COVID-19 patients. Br J Anaesth. 2021 Mar;126(3):590-598. doi: 10.1016/j.bja.2020.12.010. Epub 2020 Dec 9. PMID 33422287
- [Background] Actilyse powder and solvent SmPC 12/09/2021, NIPN: https://ogyei.gov.hu/gyogyszeradatbazis.